CLINICAL TRIAL: NCT02509689
Title: Feasibility Study of a Novel Neurofeedback Technology (GZNT) for Persistent Post-Concussive Symptoms in Soldiers
Brief Title: Neurofeedback Technology (GZNT) for Persistent Post-Concussive Symptoms in Soldiers
Acronym: GZNT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Defense and Veterans Brain Injury Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W91YTZ-13-P-0703
Record Dates: First submitted 2015-05-13; First posted 2015-07-28 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Traumatic Brain Injury
Keywords: mTBI; cognition disorders; post-concussive syndrome; neuroplasticity; EEG; biofeedback; stress disorder/post-traumatic; depression
MeSH Terms: conditions — Brain Injuries, Traumatic; Cognition Disorders; Post-Concussion Syndrome; Combat Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): The experimental intervention in this study, Global Z-Score Neurofeedback Training, is a non-pharmacological EEG Biofeedback training process using a specific new technology that allows for the training to be semi-automated and to train based on referencing EEG activity in 19 sites on the scalp, whilst comparing in real time to a database of non-clinical normative EEG data. Subjects will be scheduled to receive 20 treatment sessions of GZNT over a six-week period, aiming for four treatment visits per week, but allowing for some missed appointments due to holidays and duty obligations.
  Training will be conducted for a continuous time which will begin at 10 minutes in the first session, and progress to a maximum of 30 minutes by the sixth or seventh session, and then remain at 30 minutes of training per session for the remainder of the sessions.
  Interventions: Behavioral: Global Z-Score Neurofeedback Training

INTERVENTIONS:
Behavioral: Global Z-Score Neurofeedback Training — The experimental intervention in this study, Global Z-Score Neurofeedback Training, is a non-pharmacological EEG Biofeedback training process using a specific new technology that allows for the training to be semi-automated and to train based on referencing EEG activity in 19 sites on the scalp, whilst comparing in real time to a database of non-clinical normative EEG data. Subjects will be scheduled to receive 20 treatment sessions of GZNT over a six-week period, aiming for four treatment visits per week, but allowing for some missed appointments due to holidays and duty obligations.
  Training will be conducted for a continuous time which will begin at 10 minutes in the first session, and progress to a maximum of 30 minutes by the sixth or seventh session, and then remain at 30 minutes of training per session for the remainder of the sessions.

SUMMARY:
A new technology called Global Z-Score Neurofeedback Technology (GZNT) has been identified that can overcome an existing barrier to the use of neurofeedback as a treatment technique in a military setting. Neurofeedback, or EEG Biofeedback, is a form of biofeedback that uses the brain's own electrical activity as the training parameter. With sufficient practice, the brain can learn to change its own activity through finely tuned feedback using computerized sounds, graphs and animations. Previous attempts at using neurofeedback as a treatment modality have been subject to a lack of standardization and have required significant expertise on the part of the provider. This new GZNT technology allows neurofeedback to be administered in a standardized and semi-automated fashion, which, if effective, will represent a significant advance toward providing this promising treatment modality to Service Members in a military or VA setting. This study will determine feasibility and preliminary evidence of efficacy for this neurofeedback technology in a pilot study of soldiers with medical issues associated with Traumatic Brain Injury (TBI). GZNT technology has the potential to provide a cost-efficient, non-invasive/non-pharmacological approach to recovery from impact and/or blast-induced brain injury, and holds promise to simultaneously address emotional symptoms that are often a part of the post-concussion symptom picture.

DETAILED DESCRIPTION:
Research Design: This will be a single group design, treatment effect and feasibility study to demonstrate GZNT technology, examining electrocortical changes, and comparing emotional/vocational functioning, and post concussive symptoms before and after intensive GZNT treatment, and at three months follow-up. Up to 50 subjects with a history of traumatic brain injury and persistent cognitive and emotional symptoms will be enrolled following screening and baseline evaluation. Resting and event-related EEG (electroencephalograph) recordings, a physiological stress evaluation, neuropsychological tests, self-report symptom scales, and psychosocial/vocational functioning measures will be performed at each evaluation. All subjects will receive the study treatment intervention. Subjects will be scheduled to receive twenty treatment sessions of GZNT over a six week period, but will be counted as having completed treatment if they attend fifteen or more sessions. At least twenty-five subjects will need to complete treatment to meet statistical requirements for the study hypotheses.

Primary outcome measures will include electrocortical indices under resting and mental task states and will evaluate the degree of neuro-physiological and cortical functional connectivity change following treatment as a proxy measure for neuroplastic response to the GZNT training. Secondary outcomes will include physiological stress response (as an objective measure of emotional regulation), neuropsychological test performance (as an objective measure of cognition), and self-reported symptom and emotional well-being measures. Feasibility outcomes will include number of visits completed within the six weeks, number and reason for drop-outs, adverse event profiles, and patient satisfaction questionnaires.

Methodology/Technical: For this pilot study, the investigators will require twenty-five patients to complete the study. The investigators will therefore recruit as many as are necessary to achieve this goal, to a maximum of 50 patients. However, since this is a feasibility study, the dropout rate and reasons for drop outs will be monitored and reported. Completion of a minimum of fifteen study treatment visits will satisfy requirements for "study completion." (This is based on clinical experience data with this technology.) Therefore, only those who complete fourteen or fewer sessions within the six week study treatment time window will be counted as drop outs. The planned total number of study sessions for the study will be twenty. Data analysis will be carried out on pre and post metrics for the group who completed the trial, and secondary analyses will be carried out on all subjects using an intention-to-treat paradigm, to evaluate feasibility, and acceptance of this intervention.

Subjects will be recruited from the Warrior Recovery Center, the Soldier Readiness Center, and Evans Army Hospital Primary Care Clinics. Subjects will be pre-screened by signing an initial consent and completing a preliminary set of self-report forms, followed by a review of medical records in order to determine eligibility. Following eligibility determination, full consent discussion will be held, and baseline evaluations will be completed and study visits scheduled.

For this pilot efficacy/feasibility study, all study subjects will receive the study treatment intervention. Dose exposure will begin at 10 minutes of GZNT at the first session and progress to a maximum of thirty minutes of training by the sixth or seventh visit, and continue at thirty minutes per visit for the remainder of the study.

ELIGIBILITY:
Inclusion Criteria:

* Mild to Moderate Traumatic brain injury patients at least three months and not more than 5 years post-injury with recovery to a Rancho los Amigos level of seven or eight (alert and oriented);
* Brain injury documented in the medical record by a history of an injury event and at least one of the following:

  * loss of consciousness of any duration after the injury event;
  * post-traumatic amnesia after the injury event;
  * alteration in mental status (dazed/confused) after the injury event;
  * physical evidence of brain trauma (MRI/CT hemorrhage/contusion);
* Persistent symptoms thought to be related to or co morbid with the brain injury event, to include two or more complaints related to problems with attention, memory, concentration, speed of processing, judgment, executive control, depression, anxiety, agitation, irritability, impulsivity, or aggression, headaches, and sleep disturbance;
* Evidence of emotional problems as defined by scores on the Post-Traumatic Stress Disorder Checklist, Military version (PCL-M) of 33 or more, or 9 or more on the Patient Health Questionnaire (PHQ-9);
* Military or Veteran beneficiary;
* Males and females aged 18-50.

Exclusion Criteria:

* Current/prior (last six months) unstable medical or psychiatric condition that could confound the effect of the TBI event on brain function (e.g. clear anoxic episode, cardiac arrest, current uncontrolled diabetes, psychosis)
* A previous history of severe TBI prior to the current injury;
* Current (last three months) active suicidal or homicidal ideation or intent;
* Current (last month) drug/alcohol abuse or dependence as determined by clinical assessment in addition to the AUDIT-C screening tool. Patients with problem drinking as defined by a score of 6 or higher on the AUDIT-C will not be eligible to participate due to concerns regarding the neurotoxic effects of alcohol following TBI. Those with scores of 4 or 5 will be counseled to reduce their intake of alcohol during the time course of the study, and a clinical determination will be made by the PI or Sub-I as to whether they can be included in the study.
* Use of certain medications due to potential interference with assessments and treatment response: benzodiazepines - excluded; narcotic analgesics - allowed only if occasional use, and not within 24 hrs of any evaluation or treatment session; nootropic medications - excluded.
* Participation in a concurrent drug or treatment trial;
* Any physical impairment that prevents the patient from being able to complete the assessment or treatment tasks (including sensory functions) or failure on effort measures at baseline evaluation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Altered Electrocortical Patterns | 3 months post treatment
  EEG measures - Global Z-Score metric for 5 variables in 4 frequency bands - measure std diff within subject and for group

SECONDARY OUTCOMES:
Effects on Attention | 3 months post treatment
  Event-Related Potentials, Event-Related DeSynchronization patterns, and Behavioral Response Data from Attention Network Task
Effects on Memory | 3 months post treatment
  WAIS-IV Letter Number Sequencing, HVLT-R (auditory), BVMT-R (visual), WMS-IV Logical Memory test.

CONTACTS AND LOCATIONS:
Overall Officials: Renee M Pazdan, MD, Principal Investigator — The Defense and Veterans Brain Injury Center
Locations (1):
- Warrior Recovery Center, Bldg 1040, Fort Carson, Colorado, United States

REFERENCES:
- [Result] Hershaw JN, Hill-Pearson CA, Arango JI, Souvignier AR, Pazdan RM. Semi-Automated Neurofeedback Therapy for Persistent Postconcussive Symptoms in a Military Clinical Setting: A Feasibility Study. Mil Med. 2020 Mar 2;185(3-4):e457-e465. doi: 10.1093/milmed/usz335. PMID 31603218
- [Result] Hershaw J, Hill-Pearson CA, Arango JI, Souvignier AR, Pazdan RM. Changes in attentional processing following neurofeedback in patients with persistent post-concussive symptoms: a pilot study. Brain Inj. 2020 Dec 5;34(13-14):1723-1731. doi: 10.1080/02699052.2020.1812720. Epub 2020 Nov 16. PMID 33196305
- [Result] Hershaw JN, Hill-Pearson CA. Changes in EEG Activity Following Live Z-Score Training Predict Changes in Persistent Post-concussive Symptoms: An Exploratory Analysis. Front Neurol. 2022 Mar 21;13:714913. doi: 10.3389/fneur.2022.714913. eCollection 2022. PMID 35392637
- See also: Changes in EEG Activity Following Live Z-Score Training Predict Changes in Persistent Post-concussive Symptoms: An Exploratory Analysis — http://journal.frontiersin.org/article/10.3389/fneur.2022.714913/full?&utm_source=Email_to_authors_&utm_medium=Email&utm_content=T1_11.5e1_author&utm_campaign=Email_publication&field=&journalName=Frontiers_in_Neurology&id=